CLINICAL TRIAL: NCT05944809
Title: A Prospective Phase II Study of Prophylactic TPO Combined with Bone Marrow-sparing Intensity-modulated Radiotherapy to Reduce Platelet Inhibition in Patients with Esophageal Cancer Undergoing Concurrent Chemoradiotherapy
Brief Title: The Effect of Prophylactic TPO Combined with BMS-IMRT to Esophageal Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: JIANYANG WANG (Other)
Collaborators: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor-Investigator, JIANYANG WANG, Principal Investigator, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Organization: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NCC2818
Record Dates: First submitted 2023-06-02; First posted 2023-07-13 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Esophageal Cancer; Intensity-modulated Radiation Therapy; Concurrent Chemoradiotherapy; Thrombocytopenia
MeSH Terms: conditions — Esophageal Neoplasms; Thrombocytopenia | interventions — Chemoradiotherapy

STUDY DESIGN:
Intervention Model Description: All patients are planned to receive concurrent BMS thoracic radiotherapy (>45Gy, 1.8Gy per fraction), chemotherapy (five cycles of weekly intravenous paclitaxel [50 mg/m²] and cisplatin/nedaplatin [25 mg/m²], or two cycles of intravenous paclitaxel [135-175 mg/m²] and cisplatin/nedaplatin [80 mg/m²]) , and rhTPO，15000U ih. qw(during the radiotherapy)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- prophylactic TPO (Experimental): Prophylactic TPO combined with BMS-IMRT in the esophageal cancer patients undergoing concurrent chemoradiotherapy
  Interventions: Drug: rhTPO

INTERVENTIONS:
Drug: rhTPO — Standard treatment options:
  Radiotherapy: 95% planning target volume （planning target volume，PTV） ≥45Gy(without simultaneous boost).
  Concurrent chemotherapy:
  Weekly regimen: paclitaxel 50mg/m2 d1, nedaplatin/cisplatin 25 mg/m2d1, a total of 5 cycles.
  Three weeks regimen: paclitaxel 135-175mg/m2 d1, nedaplatin/cisplatin 80mg/m2, a total of 2 cycles.
  The active bone marrow was determined by magnetic resonance（magnetic resonance，MR）, and the dose limits are: V5<95%,V10<85%,V20<60%，V30<40%；95%PTV>45Gy.
  rhTPO，15000U ih. qw(during the radiotherapy course)
  Other Names: BMS-IMRT; concurrent chemoradiotherapy

SUMMARY:
The goal of this interventional study is to explore the protective effect of prophylactic TPO combined with bone marrow sparing (BMS)-IMRT in patients with esophageal cancer undergoing concurrent chemoradiotherapy. The main purpose is to reduce the incidence of all grades of thrombocytopenia from 35% to less than 10% by the intervention of study.

Participants will initiate concurrent chemoradiotherapy within 2 weeks after enrollment,and they will receive subcutaneous injection of recombinant human thrombopoietin (rhTPO) 15000U once a week during the radiotherapy.

DETAILED DESCRIPTION:
Concurrent chemoradiotherapy (CRT) is one of the standard treatments to the patients who initiate neoadjuvant chemoradiotherapy or radical radiotherapy. Previous large phase III trials of preoperative concurrent chemoradiotherapy and definitive chemoradiotherapy (Dt 40-60Gy) in esophageal cancer have shown rates of platelet inhibition (grade 1-4) of 25-54%. Concurrent chemotherapy has been associated with a significant increase in acute hematologic toxicity (HT) associated with radiation therapy, increasing the risk of infections, blood transfusions, colony-stimulating factors, and length of hospital stay. More importantly, severe myelosuppression also delays or interrupts the delivery of chemotherapy and radiotherapy, potentially reducing efficacy. In addition, the efficacy of locally advanced patients is still not optimistic, and the intensity of treatment may need to be increased. Therefore, if hematologic toxicity can be reduced, it may lead to more intensive concurrent chemoradiotherapy in the hope of further improving the efficacy.

Intensity-modulated radiation therapy (IMRT) has an absolute advantage over conventional radiotherapy in increasing the dose to the target volume and reducing the dose to normal tissues. Previous studies have shown a significant association between the volume of 10Gy (V10) and the volume received 20Gy (V20) of the pelvic and lumbosacral bone marrow and the development of acute HT when pelvic tumors are treated with IMRT. Thus, reducing the volume of bone marrow receiving low-dose radiotherapy may reduce the occurrence and severity of HT. Therefore, using the dosimetric advantages of IMRT, quantitative study of BMS-IMRT to reduce the toxic effects of concurrent chemoradiotherapy is a research hotspot at present.

Thrombopoietin (TPO) promotes the proliferation and survival of hematopoietic stem cells and all hematopoietic progenitor cells, accelerates the entry of stem cells into the cell cycle, and subsequently promotes the mitosis and polyploidy formation of megakaryocytes, increases the volume and number of megakaryocytes, and works with other cytokines to regulate megakaryocyte maturation. It is a commonly used drug for the treatment of thrombocytopenia in clinic.

The aim of this study is to explore the protective effect of prophylactic use of TPO on platelet inhibition in concurrent chemoradiotherapy using BMS-IMRT for esophageal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years and less than or equal to 75 years
* Histopathologically confirmed esophageal squamous/adenocarcinoma, clinical stage I-IV A (according to the 7th edition of AJCC（American Joint Committee on Cancer） 2010; Concurrent chemoradiotherapy (≥45Gy) was planned (regardless of whether the patient had received induction adjuvant chemotherapy).
* Karnofsky performance status score ≥80 ·;
* Life expectancy >6 months;
* Meet the following laboratory diagnostic criteria:

Hemoglobin ≥120g/L, white blood cell ≥4.0×109/L, Neutrophil ≥2.0×109/L, platelet ≥100×109/L;

* Participators had not used granulocyte colony-stimulating factor and thrombopoietin within 3 weeks before enrollment.

Exclusion Criteria:

* A history of malignancy at other sites, excluding curable non-melanotic skin cancer and cervical carcinoma in situ;
* Previous radiotherapy to the chest;
* Patients with existing or suspected (thoracolumbar and pelvic) bone marrow or bone metastases, or a history of bone trauma in this region within 4 weeks;
* Allergy to Gadolinium-based contrast agent;
* Patients with active infection, or combined with rheumatic immune disease, long-term chronic infection, acute infection, etc., so that the body is in an inflammatory state; Blood system diseases with hematopoietic dysfunction;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2023-07-20 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
The highest grade of thrombocytopenia (CTCAE 4.0) during the radiotherapy and 1 month after the radiotherapy. | From start of radiotherapy and 1 month after the radiotherapy.
  For esophageal cancer patients, Grade 1-4 thrombocytopenia is considered as endpoints.

SECONDARY OUTCOMES:
Physical dosimetry of active bone marrow in BMS radiotherapy plan. | The first day of radiotherapy.
  Low dose volume, the volume of active BM receiving 5,10,20,30 and 40 Gy
Conformity of BMS IMRT/VMAT (Volumetric Modulated Arc Therapy，VMAT) plan | The first day of radiotherapy.
  Conformity Index (CI）was used to evaluate the conformity of IMRT/VMAT plan.
Homogeneity of IMRT/VMAT (Volumetric Modulated Arc Therapy，VMAT) plan | The first day of radiotherapy.
  Homogeneity Index (HI) was used to evaluate the homogeneity of BMS IMRT plan.
The highest grade of leukopenia, neutropenia,anemia (CTCAE 4.0) during the radiotherapy and 1 month after the radiotherapy. | From start of radiotherapy and 1 month after the radiotherapy.
  For esophageal cancer patients, Grade 1-4 leukopenia, neutropenia and anemia are considered as endpoints.

CONTACTS AND LOCATIONS:
Overall Officials: Jianyang Wang, MD, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences & Peking Union Medical College
Locations (1):
- Department of Radiation Oncology, Cancer Institute and Hospital, Chinese Academy of Medical Sciences & Peking Union Medical College, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van Hagen P, Hulshof MC, van Lanschot JJ, Steyerberg EW, van Berge Henegouwen MI, Wijnhoven BP, Richel DJ, Nieuwenhuijzen GA, Hospers GA, Bonenkamp JJ, Cuesta MA, Blaisse RJ, Busch OR, ten Kate FJ, Creemers GJ, Punt CJ, Plukker JT, Verheul HM, Spillenaar Bilgen EJ, van Dekken H, van der Sangen MJ, Rozema T, Biermann K, Beukema JC, Piet AH, van Rij CM, Reinders JG, Tilanus HW, van der Gaast A; CROSS Group. Preoperative chemoradiotherapy for esophageal or junctional cancer. N Engl J Med. 2012 May 31;366(22):2074-84. doi: 10.1056/NEJMoa1112088. PMID 22646630
- [Background] Yang H, Liu H, Chen Y, Zhu C, Fang W, Yu Z, Mao W, Xiang J, Han Y, Chen Z, Yang H, Wang J, Pang Q, Zheng X, Yang H, Li T, Lordick F, D'Journo XB, Cerfolio RJ, Korst RJ, Novoa NM, Swanson SJ, Brunelli A, Ismail M, Fernando HC, Zhang X, Li Q, Wang G, Chen B, Mao T, Kong M, Guo X, Lin T, Liu M, Fu J; AME Thoracic Surgery Collaborative Group. Neoadjuvant Chemoradiotherapy Followed by Surgery Versus Surgery Alone for Locally Advanced Squamous Cell Carcinoma of the Esophagus (NEOCRTEC5010): A Phase III Multicenter, Randomized, Open-Label Clinical Trial. J Clin Oncol. 2018 Sep 20;36(27):2796-2803. doi: 10.1200/JCO.2018.79.1483. Epub 2018 Aug 8. PMID 30089078
- [Background] Chen Y, Ye J, Zhu Z, Zhao W, Zhou J, Wu C, Tang H, Fan M, Li L, Lin Q, Xia Y, Li Y, Li J, Jia H, Lu S, Zhang Z, Zhao K. Comparing Paclitaxel Plus Fluorouracil Versus Cisplatin Plus Fluorouracil in Chemoradiotherapy for Locally Advanced Esophageal Squamous Cell Cancer: A Randomized, Multicenter, Phase III Clinical Trial. J Clin Oncol. 2019 Jul 10;37(20):1695-1703. doi: 10.1200/JCO.18.02122. Epub 2019 Mar 28. PMID 30920880
- [Background] Ji Y, Du X, Zhu W, Yang Y, Ma J, Zhang L, Li J, Tao H, Xia J, Yang H, Huang J, Bao Y, Du D, Liu D, Wang X, Li C, Yang X, Zeng M, Liu Z, Zheng W, Pu J, Chen J, Hu W, Li P, Wang J, Xu Y, Zheng X, Chen J, Wang W, Tao G, Cai J, Zhao J, Zhu J, Jiang M, Yan Y, Xu G, Bu S, Song B, Xie K, Huang S, Zheng Y, Sheng L, Lai X, Chen Y, Cheng L, Hu X, Ji W, Fang M, Kong Y, Yu X, Li H, Li R, Shi L, Shen W, Zhu C, Lv J, Huang R, He H, Chen M. Efficacy of Concurrent Chemoradiotherapy With S-1 vs Radiotherapy Alone for Older Patients With Esophageal Cancer: A Multicenter Randomized Phase 3 Clinical Trial. JAMA Oncol. 2021 Oct 1;7(10):1459-1466. doi: 10.1001/jamaoncol.2021.2705. PMID 34351356
- [Background] Li C, Tan L, Liu X, Wang X, Zhou Z, Chen D, Feng Q, Liang J, Lv J, Wang X, Bi N, Deng L, Wang W, Zhang T, Ni W, Chang X, Han W, Gao L, Wang S, Xiao Z. Concurrent chemoradiotherapy versus radiotherapy alone for patients with locally advanced esophageal squamous cell carcinoma in the era of intensity modulated radiotherapy: a propensity score-matched analysis. Thorac Cancer. 2021 Jun;12(12):1831-1840. doi: 10.1111/1759-7714.13971. Epub 2021 May 5. PMID 33949784
- [Background] Liu Y, Zheng Z, Li M, Zhang Y, Zhao F, Gong H, Lin H, Huang W, Chen X, Xu Z, Li X, Liu W, Cui Y, Zheng A, Li B. Comparison of concurrent chemoradiotherapy with radiotherapy alone for locally advanced esophageal squamous cell cancer in elderly patients: A randomized, multicenter, phase II clinical trial. Int J Cancer. 2022 Aug 15;151(4):607-615. doi: 10.1002/ijc.34030. Epub 2022 Apr 27. PMID 35419831
- [Background] Abu-Rustum NR, Lee S, Correa A, Massad LS. Compliance with and acute hematologic toxic effects of chemoradiation in indigent women with cervical cancer. Gynecol Oncol. 2001 Apr;81(1):88-91. doi: 10.1006/gyno.2000.6109. PMID 11277656
- [Background] Green JA, Kirwan JM, Tierney JF, Symonds P, Fresco L, Collingwood M, Williams CJ. Survival and recurrence after concomitant chemotherapy and radiotherapy for cancer of the uterine cervix: a systematic review and meta-analysis. Lancet. 2001 Sep 8;358(9284):781-6. doi: 10.1016/S0140-6736(01)05965-7. PMID 11564482
- [Background] Torres MA, Jhingran A, Thames HD Jr, Levenback CF, Bodurka DC, Ramondetta LM, Eifel PJ. Comparison of treatment tolerance and outcomes in patients with cervical cancer treated with concurrent chemoradiotherapy in a prospective randomized trial or with standard treatment. Int J Radiat Oncol Biol Phys. 2008 Jan 1;70(1):118-25. doi: 10.1016/j.ijrobp.2007.05.028. Epub 2007 Sep 14. PMID 17869451
- [Background] Rose PG, Bundy BN, Watkins EB, Thigpen JT, Deppe G, Maiman MA, Clarke-Pearson DL, Insalaco S. Concurrent cisplatin-based radiotherapy and chemotherapy for locally advanced cervical cancer. N Engl J Med. 1999 Apr 15;340(15):1144-53. doi: 10.1056/NEJM199904153401502. PMID 10202165
- [Background] Nugent EK, Case AS, Hoff JT, Zighelboim I, DeWitt LL, Trinkhaus K, Mutch DG, Thaker PH, Massad LS, Rader JS. Chemoradiation in locally advanced cervical carcinoma: an analysis of cisplatin dosing and other clinical prognostic factors. Gynecol Oncol. 2010 Mar;116(3):438-41. doi: 10.1016/j.ygyno.2009.09.045. Epub 2009 Nov 5. PMID 19896180
- [Background] Brixey CJ, Roeske JC, Lujan AE, Yamada SD, Rotmensch J, Mundt AJ. Impact of intensity-modulated radiotherapy on acute hematologic toxicity in women with gynecologic malignancies. Int J Radiat Oncol Biol Phys. 2002 Dec 1;54(5):1388-96. doi: 10.1016/s0360-3016(02)03801-4. PMID 12459361
- [Background] Roeske JC, Lujan A, Rotmensch J, Waggoner SE, Yamada D, Mundt AJ. Intensity-modulated whole pelvic radiation therapy in patients with gynecologic malignancies. Int J Radiat Oncol Biol Phys. 2000 Dec 1;48(5):1613-21. doi: 10.1016/s0360-3016(00)00771-9. PMID 11121668
- [Background] Mundt AJ, Lujan AE, Rotmensch J, Waggoner SE, Yamada SD, Fleming G, Roeske JC. Intensity-modulated whole pelvic radiotherapy in women with gynecologic malignancies. Int J Radiat Oncol Biol Phys. 2002 Apr 1;52(5):1330-7. doi: 10.1016/s0360-3016(01)02785-7. PMID 11955746
- [Background] Gershkevitsh E, Rosenberg I, Dearnaley DP, Trott KR. Bone marrow doses and leukaemia risk in radiotherapy of prostate cancer. Radiother Oncol. 1999 Dec;53(3):189-97. doi: 10.1016/s0167-8140(99)00145-0. PMID 10660197
- [Background] Mell LK, Kochanski JD, Roeske JC, Haslam JJ, Mehta N, Yamada SD, Hurteau JA, Collins YC, Lengyel E, Mundt AJ. Dosimetric predictors of acute hematologic toxicity in cervical cancer patients treated with concurrent cisplatin and intensity-modulated pelvic radiotherapy. Int J Radiat Oncol Biol Phys. 2006 Dec 1;66(5):1356-65. doi: 10.1016/j.ijrobp.2006.03.018. Epub 2006 Jun 6. PMID 16757127
- [Background] Mell LK, Schomas DA, Salama JK, Devisetty K, Aydogan B, Miller RC, Jani AB, Kindler HL, Mundt AJ, Roeske JC, Chmura SJ. Association between bone marrow dosimetric parameters and acute hematologic toxicity in anal cancer patients treated with concurrent chemotherapy and intensity-modulated radiotherapy. Int J Radiat Oncol Biol Phys. 2008 Apr 1;70(5):1431-7. doi: 10.1016/j.ijrobp.2007.08.074. Epub 2007 Nov 8. PMID 17996390
- [Background] Lhomme C, Fumoleau P, Fargeot P, Krakowski Y, Dieras V, Chauvergne J, Vennin P, Rebattu P, Roche H, Misset JL, Lentz MA, Van Glabbeke M, Matthieu-Boue A, Mignard D, Chevallier B. Results of a European Organization for Research and Treatment of Cancer/Early Clinical Studies Group phase II trial of first-line irinotecan in patients with advanced or recurrent squamous cell carcinoma of the cervix. J Clin Oncol. 1999 Oct;17(10):3136-42. doi: 10.1200/JCO.1999.17.10.3136. PMID 10506610
- [Background] Curtin JP, Blessing JA, Webster KD, Rose PG, Mayer AR, Fowler WC Jr, Malfetano JH, Alvarez RD. Paclitaxel, an active agent in nonsquamous carcinomas of the uterine cervix: a Gynecologic Oncology Group Study. J Clin Oncol. 2001 Mar 1;19(5):1275-8. doi: 10.1200/JCO.2001.19.5.1275. PMID 11230468
- [Background] Kaushansky K. Thrombopoietin. N Engl J Med. 1998 Sep 10;339(11):746-54. doi: 10.1056/NEJM199809103391107. No abstract available. PMID 9731092